CLINICAL TRIAL: NCT01302730
Title: A Self-Administered Questionnaire for Early Detection of Axial Spondyloarthritis
Brief Title: Ankylosing Spondylitis and Spondyloarthritis Evaluation Tool Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); Oregon Health and Science University (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Eswar Krishnan, ASSISTANT PROFESSOR, Stanford University
Other Study IDs: STANIRB-20278
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Ankylosing Spondylitis; Spondylarthritis
Keywords: ankylosing spondylitis; spondylarthritis; inflammatory back pain; seronegative
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to test whether a new instrument (questionnaire) is useful for identifying patients with ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to rheumatologist office will be potentially eligible.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Physician diagnosis of Ankylosing Spondylitis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eswar Krishnan, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States